CLINICAL TRIAL: NCT04348825
Title: Effects of ECT in Treatment of Major Depression: A Prospective Neuroradiological Study of Acute and Longitudinal Effects on Brain Structure and Function
Brief Title: Electroconvulsive Therapy and Neuroradiology
Acronym: ECTMRI
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Other Study IDs: 2013/1032
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2020-05

CONDITIONS: Depression; Electroconvulsive Therapy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients, depression: Patients who receive ECT as part of clinical care
  Interventions: Device: Electroconvulsive therapy
- Healthy: Healthy controls who do not receive ECT but otherwise the same assessments.
- Patients, atrial fibrilation: Patients who receive Electro Cardio Version (ECV) due to Atrial Fibrilation

INTERVENTIONS:
Device: Electroconvulsive therapy
  Groups: Patients, depression

SUMMARY:
The study will apply state of the art radiology through advanced magnetic resonance imaging (MRI) techniques to investigate structural and functional brain effects of ECT.

DETAILED DESCRIPTION:
As a multi-disciplinary collaboration, imaging findings will be correlated to psychiatric response parameters, neuropsychological functioning as well as neurochemical and genetic biomarkers that can elucidate the underlying mechanisms. The aim is to document both treatment effects and potential harmful effects of ECT.

Sample: n = 40 patients in a major depressive episode (bipolar and major depressive disorder). Two control groups with n = 15 in each group: age and gender matched healthy volunteers not receiving ECT and patients undergoing electrical cardioversion (ECV) for atrial fibrillation (AF). Observation time: six months.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age > 18) referred to the ECT-unit and accepted for treatment because of moderate and severe depression,
* fulfilling the criteria for the following ICD-10 diagnoses: F31.3 and F31.4; F32.1 and F32.2 and F32.3; F33.1 and F33.2 and F33.3.
* symptom intensity must be verified by a score ≥ 25 on the Montgomery and Åsberg Depression Rating Scale (MADRS).

Exclusion Criteria:

* ECT treatment within the last 12 months.
* Pregnancy.
* Patients unable to give written informed consent (according to the responsible clinician or ECT responsible).
* Patients who cannot participate in the MRI scanning because of contraindications to MRI.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Forty patients accepted for ECT at Haukeland University Hospital will be included.
  Control groups: A group of patients undergoing Electrocardioversion (ECV) for atrial fibrilation (AF) (controls 1) and healthy controls undergoing the same investigations as the ECT patient group, but not receiving ECT or anesthesia (controls 2).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Magnetic Resonance Imaging (MRI) derived parameters | Before (baseline), during, after (typically 1-2 weeks after last ECT) and at follow up (6 months after treatment)
  MRI of the brain is segmented into Regions of Interest by automated processing pipelines
Changes from baseline in Depression ratings | Before (baseline), during, after (typically 1-2 weeks after last ECT) and at follow up (6 months after treatment)
  Symptoms scores on Montgomery-Åsberg Depression Rating Scale (MADRS)

SECONDARY OUTCOMES:
Changes from baseline in Neurocognitive functioning | Before (baseline), after (typically 1-2 weeks after last ECT) and at follow up (6 months after treatment)
  Neurocognitive assessments

CONTACTS AND LOCATIONS:
Overall Officials: Ketil J Ødegaard, PhD, Principal Investigator — Haukeland University Hospital

REFERENCES:
- [Background] Oltedal L, Kessler U, Ersland L, Gruner R, Andreassen OA, Haavik J, Hoff PI, Hammar A, Dale AM, Hugdahl K, Oedegaard KJ. Effects of ECT in treatment of depression: study protocol for a prospective neuroradiological study of acute and longitudinal effects on brain structure and function. BMC Psychiatry. 2015 May 1;15:94. doi: 10.1186/s12888-015-0477-y. PMID 25927716
- [Derived] Hammar A, Ronold EH, Spurkeland MA, Ueland R, Kessler U, Oedegaard KJ, Oltedal L. Improvement of persistent impairments in executive functions and attention following electroconvulsive therapy in a case control longitudinal follow up study. BMC Psychiatry. 2024 Nov 20;24(1):832. doi: 10.1186/s12888-024-06270-5. PMID 39567961
- [Derived] Blomberg MO, Semkovska M, Kessler U, Erchinger VJ, Oedegaard KJ, Oltedal L, Hammar A. A Longitudinal Comparison Between Depressed Patients Receiving Electroconvulsive Therapy and Healthy Controls on Specific Memory Functions. Prim Care Companion CNS Disord. 2020 May 14;22(3):19m02547. doi: 10.4088/PCC.19m02547. PMID 32408397